CLINICAL TRIAL: NCT02195297
Title: Clinical and Instrumental Evaluation of the Activity of a Pharmacological "Anticellulitis" Product vs. a Reference Product on the Market: Comparison Within Subjects (Double Blind Study)
Brief Title: Evaluation of the Activity of a Pharmacological "Anticellulitis" Product vs. a Reference Product on the Market
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: E1513
Record Dates: First submitted 2014-07-10; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: cellulitis; anticellulitis
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ANTICELLULITE GMG GIULIANI (Active Comparator): Each included subject applied ANTICELLULITE GMG GIULIANI mono-laterally (on the left or on right side according to a previously defined randomization list) once a day, at evening, for an uninterrupted period of 4 weeks.
  Interventions: Other: ANTICELLULITE GMG GIULIANI Cream and SOMATOLINE Cream
- SOMATOLINE (Active Comparator): Each included subject applied SOMATOLINE CREAM mono-laterally (on the left or on right side according to a previously defined randomization list) once a day, at evening, for an uninterrupted period of 4 weeks.
  Interventions: Other: ANTICELLULITE GMG GIULIANI Cream and SOMATOLINE Cream

INTERVENTIONS:
Other: ANTICELLULITE GMG GIULIANI Cream and SOMATOLINE Cream — Products application: mono-laterally, once a day at evening (4 doses from each dispenser for the first 2 day-treatment and 2 doses for the following days)

SUMMARY:
Aim of this study was to evaluate by clinical, morphometric and non invasive instrumental evaluations the activity of an "anticellulitis" cosmetic product vs a reference product of the market (comparison within subjects), applied once a day, for an uninterrupted period of 4 weeks, on 22 female healthy volunteers with low/moderate oedematous - fibrosclerotic lipodystrophy on the thighs.

It was also aim of the study to evaluate cosmetic acceptability by the volunteers and products efficacy and tolerance both by investigator and volunteers.

ELIGIBILITY:
Inclusion Criteria:

* female volunteers
* volunteers aged more than 18 years old
* volunteers with low/moderate oedematous - fibrosclerotic lipodystrophy on the thighs
* volunteers with no weight variation (± 1.5 kg) during the last month preceding the study inclusion
* volunteers with regular menstrual cycle (28-32 days) or in menopause from at least 2 years
* volunteers who are giving a written informed consent.

Exclusion Criteria:

* pregnancy
* lactation
* smoke (admitted 10 cigarettes/day)
* assumption of alcoholic drinks/wine/beer (admitted up to 125 ml for meal)
* oral contraceptive/replacement therapy started less than 1 year ago
* alimentary diet
* change in the normal habits in the last month (unusual physical activity)
* use of any product or weight-loss treatment (manual or instrumental massage) on skin test areas during the last month
* use of any drug able to cause a weight body variation
* presence of clinically important vascular disorders
* insufficient adhesion to the study protocol and to the treatment
* participation in a similar study during the previous month
* dermatological disease
* clinical and significant skin condition on the test area (e.g. lesions, scars, malformations)
* suspect thyroid disfunction
* thyroid disorders/diseases
* other endocrine diseases as diabetes, metabolic disorders etc.
* hepatic, renal or cardiac disorder
* cancer
* topical drugs or surgical procedure on the test areas during the previous 3 months
* systemic corticosteroids
* aspirin or non-steroid anti-inflammatory drugs (FANS)
* diuretic drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Morphometric evaluations: change from baseline (T2 and T4 vs. T0) | after 2 and 4 week-treatment
  All the measures were performed in standard conditions at level of the thigh (III superior, III middle and inferior), thanks to a specific electro-optical system.

SECONDARY OUTCOMES:
Ultrasonographic evaluations: change from baseline (T2 and T4 vs. T0) | after 2 and 4 week-treatment
  Ultrasonographic measurement of adipose panniculum thickness (mm) was performed at level of the external thigh (III superior) through the instrument Body Metrix™ BX 2000 (Genex).
Skin plastoelasticity: change from baseline (T2 and T4 vs. T0) | after 2 and 4 week-treatment
  Skin elasticity was measured through the instrument Dermal Torque Meter (Dia-Stron Ltd., UK). This instrument is based on the principle of the torsion given to the skin surface by a probe made of two circles that adhere to the skin through shaped adhesive tapes. The instrument measures the torsion angle (θ) during the mechanical stimulus ("torque on") and after it has ceased ("torque off"). For each of the considered curves it was measured the cutaneous rotational ratio relative to defined measured times, obtaining the parameters listed below:
  Ue: immediate extensibility ("torque on" at 0.2 sec.) Uf: final extensibility ("torque on" at 9 sec.) Uv: viscoelasticity Ur: immediate elastic recovery ("torque off" at 0.2 sec.)
Tissue dielectric constant of deep skin layers: change from baseline (T2 and T4 vs. T0) | after 2 and 4 week-treatment
  Tissue dielectric constant of deep skin layers misures non-invasively the dielectric constant of the subcutaneous fat; it is a dimensionless physical quantity and it is directly proportional to the water content in the measured tissue. The used probe corresponds to an effective measurement depth of 5 mm; the measure were performed at level of the external thigh (III superior).
Optical densitometry: change from baseline (T2 and T4 vs. T0) | after 2 and 4 week-treatment
  The measurement of the skin erythema at level of the internal area of the knee was performed by the use of an optical densitometer (X-RITE 404) allowing to quantify, on a logarithmic scale, total reflected optical density (visual=V) and the values of primary subtractive colours of reflected light: cyan(=C), magenta(=M) and yellow(=Y). Calculation of erythema index was done as follows: E.I.=logRmagenta-logRcyan, where R represents the reflectance.
Thermography evaluation: change from baseline (T2 and T4 vs. T0) | after 2 and 4 week-treatment
  Contact thermography permits visualizing, through colors, the temperatures of the areas being examined by using encapsulated liquid crystals plates; it allows to detect information about cutaneous microcirculation in normal conditions, after functional stimuli or vasoactive treatments: skin temperature grows in case of vasodilatation, increase of blood vessels, increase local metabolism and reduced in case of vasoconstriction, pathological decrease of blood vessels, decrease of local metabolism, oedema and increase of adipose tissue. A characteristic thermography aspect of legs' oedematous - fibrosclerotic lipodystrophy is represented by the typical leopard skin with large hypothermic zones. Panniculopatia evaluation follows next classification:
  0 = uniform hyperthermal image
  1. = shaded spots thermal image (hyperthermal images)
  2. = leopard spots (numerous hyperthermal images)
  3. = hypothermal black holes
  4. = uniform hypothermal image
Clinical evaluations: change from baseline (T2 and T4 vs. T0) | after 2 and 4 week-treatment
  Performed at level of the III superior, of the III middle and inferior of the thigh:
  * cellulitis visual aspect (according to a reference photographic scale) no cellulitis 0 slight dimpling on skin surface 1 dimpling and skin depressions 2 dimpling and depressed striations 3 nodules and depressed striations 4
  * cellulitis aspect to pinching ( according to a reference photographic scale) no cellulitis 0 slight dimpling on skin surface 1 dimpling and skin depressions 2 dimpling and depressed striations 3 nodules and depressed striations 4
  * pain at pinching absent 0 slight 1 medium 2 consistent 3 very consistent 4
  * firmness (internal thigh) very poor 0 poor 1 medium 2 good 3 very good 4
  * smoothness very poor 0 poor 1 medium 2 good 3 very good 4

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, Doctor, Principal Investigator — Derming SRL

REFERENCES:
- [Background] Alanen E, Lahtinen T, Nuutinen J. Penetration of electromagnetic fields of an open-ended coaxial probe between 1 MHz and 1 GHz in dielectric skin measurements. Phys Med Biol. 1999 Jul;44(7):N169-76. doi: 10.1088/0031-9155/44/7/404. PMID 10442720
- [Background] Bellisari A. Sonographic Measurement of adipose tissue. J. Diagn. Med. Sonogr., 9 (1): 11-18, 1993
- [Background] Bellisari A, Roche AF, Siervogel RM. Reliability of B-mode ultrasonic measurements of subcutaneous adipose tissue and intra-abdominal depth: comparisons with skinfold thicknesses. Int J Obes Relat Metab Disord. 1993 Aug;17(8):475-80. PMID 8401751
- [Background] Curri SB. Cellulite. Doctor dermatologia, 1: 39-52,1991.
- [Background] Curri SB. Adiposità localizzata e pannicolopatia edemato-fibrosclerotica. Sepem, Milano, 1990
- [Background] De Rigal J, Leveque JL. In vivo measurement of the stratum corneum elasticity Bioengineering and the skin 1: 13-23, 1985
- [Background] Fernay, Voltaire. The World Medical Association (1989) "World Medical Association Declaration of Helsinki", Hong-Kong.
- [Background] ICH Harmonised Tripartite Guideline - Guideline for Good Clinical Practice International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use: May (1996)
- [Background] Kiiskinen M., Nuutinen J. and Alanen E. Measurement depths of a skin-water analyzer (MoistureMeter D)Skin Res Technol, Vol 11: 292, (2005)
- [Background] Lahtinen, T., Nuutinen, J., Alanen, E. Dielectric properties of the skin In: Radio Frequency Radiation Dosimetry. Editors: B. J. Klauenberg and D. Miklavcic. Kluwer Academic Publishers, the Netherlands, (2000)
- [Background] Lahtinen T, Nuutinen J, Alanen E. Dielectric properties of the skin. Phys Med Biol. 1997 Jul;42(7):1471-2. doi: 10.1088/0031-9155/42/7/020. No abstract available. PMID 9253055
- [Background] Radic R, Nikolic V, Karner I, Kurbel S, Selthofer R. Ultrasound measurement in defining the regional distribution of subcutaneous fat tissue. Coll Antropol. 2002 Dec;26 Suppl:59-68. PMID 12674836
- [Background] Ramirez ME. Measurement of subcutaneous adipose tissue using ultrasound images. Am J Phys Anthropol. 1992 Nov;89(3):347-57. doi: 10.1002/ajpa.1330890308. PMID 1485642
- [Background] Rieger M.M., Battista G.W. Some experiences in the safety testing of cosmetics J. Soc. Cosmet. Chem. 15:161 -172, (1964)
- [Background] Sachs L Applied statistics: a handbook of techniques. Heidelberg: Springer,:536-539, (1981)
- [Background] Salter DC, McArthur HC, Crosse JE, Dickens AD. Skin mechanics measured in vivo using torsion: a new and accurate model more sensitive to age, sex and moisturizing treatment. Int J Cosmet Sci. 1993 Oct;15(5):200-18. doi: 10.1111/j.1467-2494.1993.tb00075.x. PMID 19272125
- [Background] Sparavigna A., Setaro M., Galbiati G. Osservazioni sull'elasticità della pelle Cosmesi Dermatologica 22:68-78, (1988)
- [Background] Sparavigna A., Setaro M., A new evaluation method of skin plastoelasticity in skin pharmacology and toxicology. Recent advances. Plenum Publishing Corporation, New York, London: 295-298, (1990)
- [Background] Sparavigna A., Galbiati G. La plastoelasticità cuanea: Metodi di indagine e significato clinico Chronica Dermatologica 4: 509-517, (1992)
- [Background] Sparavigna A., Setaro M. Misurazione delle propietà meccaniche della cute mediante metodi di torsione In:"Diagnostica non invasiva in dermatologia" A cura di Stefania Seidenari, EDRA Medical Publishing & New Media, Milano, Pagg. 323-328, (1998)
- [Background] Van de Vijver LPL, Boelsma E, Bausch-Goldbohm RA, Roza L Subjective skin condition and its association with objective skin measurements. Cosm Toil: 118: 45-54, (2003)
- [Background] Bayrakci Tunay V, Akbayrak T, Bakar Y, Kayihan H, Ergun N. Effects of mechanical massage, manual lymphatic drainage and connective tissue manipulation techniques on fat mass in women with cellulite. J Eur Acad Dermatol Venereol. 2010 Feb;24(2):138-42. doi: 10.1111/j.1468-3083.2009.03355.x. Epub 2009 Jul 13. PMID 19627407
- See also: Investigation center — http://www.derming.com/
- See also: Sponsor — http://www.giulianipharma.com/